CLINICAL TRIAL: NCT00947024
Title: The Effect of Food on the Bioavailability of Glipizide
Brief Title: To Demonstrate the Effect of Food on the Bioavailability of Glipizide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9301813
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glipizide

ARMS (3):
- 1 (Experimental): 10 mg Glipizide Tablet (Geneva Pharmaceutical, Inc.), Administered Immediately After a Standard Breakfast.
  Interventions: Drug: 10 mg Glipizide Tablet (Geneva Pharmaceutical, Inc.), Administered Immediately After a Standard Breakfast.
- 3 (Active Comparator): 10 mg Glucotrol Tablet (Roerig), Administered Immediately After a Standard Breakfast.
  Interventions: Drug: 10 mg Glucotrol Tablet (Roerig), Administered Immediately After a Standard Breakfast.
- 2 (Experimental): 10 mg Glipizide Tablet (Geneva Pharmaceutical, Inc.), Administered After an Overnight Fast.
  Interventions: Drug: 10 mg Glipizide Tablet (Geneva Pharmaceutical, Inc.), Administered After an Overnight Fast.

INTERVENTIONS:
Drug: 10 mg Glipizide Tablet (Geneva Pharmaceutical, Inc.), Administered Immediately After a Standard Breakfast.
  Arms: 1
Drug: 10 mg Glucotrol Tablet (Roerig), Administered Immediately After a Standard Breakfast.
  Arms: 3
Drug: 10 mg Glipizide Tablet (Geneva Pharmaceutical, Inc.), Administered After an Overnight Fast.
  Arms: 2

SUMMARY:
To demonstrate the effect of food on the bioavailability of Glipizide.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 1993-11; Primary Completion 1993-11 (Actual); Study Completion 1993-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Roger D. Anderson, M.D., Principal Investigator — Novum Pharmaceutical Research Services